CLINICAL TRIAL: NCT06114459
Title: Impact of Postoperative Skin Disinfection With Chlorhexidine on Bacterial Colonization Following Shoulder Arthroplasty Surgery: A Controlled Randomized Study
Brief Title: Impact of Postoperative Skin Disinfection With Chlorhexidine on Bacterial Colonization
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Linkoeping University (Other Government)
Responsible Party: Principal Investigator, Ida Markstrom, CORN,, Linkoeping University
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Prevention
Other Study IDs: 780727
Record Dates: First submitted 2023-10-28; First posted 2023-11-02 (Actual); Last update posted 2023-11-02 (Actual); Status verified 2023-10

CONDITIONS: Surgical Site Infection
MeSH Terms: conditions — Surgical Wound Infection | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chlorhexidine (Experimental): Postoperative disinfection
  Interventions: Drug: Sodium Chloride
- Sodium Chloride (Experimental): Postoperative disinfection
  Interventions: Drug: Sodium Chloride

INTERVENTIONS:
Drug: Sodium Chloride — Post surgery disinfection

SUMMARY:
A double-blinded, controlled study was conducted at one county hospital in Sweden. Patients were randomly assigned, skin samples were collected at four times; baseline, preoperative, after intervention and after 48 hours. Bacterial colonization were assessed.

DETAILED DESCRIPTION:
METHOD Study design

This was a double blinded, controlled, block-randomized intervention study with random allocation to Chlorhexidine- group or Sodium Chloride- group.

Sample and setting Participants was recruited at one county hospital in the southeast of Sweden from august 2019 to mars 2023. Consecutive sampling of adult patients over 18 years of age scheduled for primary elective shoulder arthroplasty surgery was approached for participation.

Intervention According to a predetermined schedule, the surgery site was either disinfected with 5 mg chlorhexidine in 70% ethanol or cleaned with sterile sodium chloride, Skin samples Skin swabs were collected on four occasions: 1. Baseline, 2. After skin disinfection, 3. Post-intervention, and 4. After 48 hours. All samples in the study were collected utilizing the eSwab system with flocked swabs Two swabs were collected on each occasion. The Pencil Eraser Swab (PES)- technique was employed (26). Swabs were gently rubbed in an oscillating motion, moving downward, and then replicating the same motion upward, repeated 15 times. For sample 1 and 2, one swab on each side of the intended incision site was collected. For samples 3 and 4, swabs were taken from each sides of the incision, positioned 1 cm away from the sutures or staples, with one swab collected on each side

ELIGIBILITY:
Inclusion Criteria: Adult patients over 18 years, scheduled for primary elective shoulder arthroplasty surgery.

Exclusion Criteria: Exclusion criteria were previous allergic reaction or perceived adverse effects of chlorhexidine, prolonged treatment with cortisone (>5 mg), antibiotic treatment within 14 days prior to scheduled surgery, skin disease or ongoing skin infection.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-08-10 (Actual); Primary Completion 2023-03-20 (Actual); Study Completion 2023-03-20 (Actual)

PRIMARY OUTCOMES:
Bacterial colonization | At 48 hours after shoulder surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Ryhov Hospital, Jönköping, Småland, Sweden

IPD SHARING:
Plan to Share IPD: No